CLINICAL TRIAL: NCT04036487
Title: Chimay Plastic Surgery Clinic, Taipei
Brief Title: Effects of General Anesthesia on Quality of Recovery After Transaxillary Endoscopic Breast Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Cheng Hung (Other)
Responsible Party: Sponsor-Investigator, Chih-Cheng Hung, Superintendent, Chimay Plastic Surgery Clinic
Organization: Chimay Plastic Surgery Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMTMU201701
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Breast Augmentation; Inhalation Anesthesia; Total Intravenous Anesthesia; Quality of Recovery
MeSH Terms: interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IH group (Experimental): Inhalation anesthesia will be given during transaxillary endoscopic breast augmentation.
  Interventions: Drug: Desflurane
- TIVA group (Active Comparator): Total intravenous anesthesia will be given during transaxillary endoscopic breast augmentation.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — Anesthesia is maintained by desflurane in an oxygen air mixture of 60/40%. If inadequate depth of anesthesia is observed, the end-expiratory concentration of desflurane would be increased.
  Arms: IH group
Drug: Propofol — Anesthesia is maintained by propofol 100-200 μg/kg/min. If inadequate depth of anesthesia is observed, the rate of propofol infusion would be increased.
  Arms: TIVA group

SUMMARY:
Among aesthetic or cosmetic surgeries, breast augmentation was the most frequently performed and the endoscopic transaxillary approach has become the preferred incision for Asian women. As breast augmentation must be performed under general anesthesia accompanied by its effects and potential complications, types of general anesthesia may affect the quality of recovery. Currently, the two most common techniques of general anesthesia are inhalation anesthesia (IH) and total intravenous anesthesia (TIVA). The effects of these types of general anesthesia on the quality of recovery have been investigated for numerous surgical procedures. However, no prior studies have analyzed different types of anesthesia used for performing transaxillary endoscopic breast augmentation. This prospective, parallel, randomized controlled study will evaluate the effects of inhalation anesthesia vs. total intravenous anesthesia on the quality of recovery in patients undergoing transaxillary endoscopic breast augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients are appropriate for undergoing transaxillary endoscopic breast augmentation
* Age between 20-65 years
* Physical Status I or II as defined by the American Society of Anesthesiologists (ASA) Physical Status Classification System

Exclusion Criteria:

* Having difficulty reading or hearing
* Diagnosed with addictive disorder
* Diagnosed with psychiatric disorder
* Physical Status III-VI as defined by the ASA Physical Status Classification System
* Presence of acute infection or inflammatory condition (e.g., fever).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Quality of recovery, postoperative day one | On the 1st postoperative day
  Quality of recovery is assessed by the 15-item Quality of Recovery (QoR-15) questionnaire. The total score of the 15-item QoR ranges from 0 to 150, and a higher score indicates a better outcome.
Quality of recovery, postoperative day two | On the 2nd postoperative day
  Quality of recovery is assessed by the 15-item Quality of Recovery (QoR-15) questionnaire. The total score of the 15-item QoR ranges from 0 to 150, and a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Chimay Plastic Surgery Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No